CLINICAL TRIAL: NCT01011608
Title: Effect of a Medical Food Supplement in Hospitalized Patients Recovering From Hip Fracture Surgery
Brief Title: Effect of a Medical Food Supplement in Hospitalized Patients Recovering From Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott Nutrition (Industry)
Responsible Party: Bobbie Swearengin, Director Clinical Research Operations, Abbott Nutrition
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BK52
Record Dates: First submitted 2009-11-10; First posted 2009-11-11 (Estimated); Last update posted 2011-04-04 (Estimated); Status verified 2010-11

CONDITIONS: Hip Fracture
MeSH Terms: conditions — Hip Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Medical Food Supplement (Experimental): Medical food supplement to be given in divided portions in morning, afternoon and evening
  Interventions: Other: Medical Food Supplement
- standard hospital food (Active Comparator): standard hospital diet
  Interventions: Other: standard hospital food

INTERVENTIONS:
Other: Medical Food Supplement — Medical Food Supplement to be given in divided portions in morning, afternoon and evening
  Arms: Medical Food Supplement
Other: standard hospital food — standard hospital diet ad. lib.
  Arms: standard hospital food

SUMMARY:
The objective of this study is to evaluate the effect of nutritional supplementation on the nutritional and clinical course of patients admitted to the hospital for hip fracture surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subject is > 45 years of age.
* Subject is a male or a non-pregnant, non-lactating female, at least 6 weeks postpartum prior to screening visit.
* Subject plans to undergo hip fracture surgery.
* Subject has anticipated length of hospital stay of at least 4 weeks. Subject is able to consume foods and beverages orally.
* Subject has admission total protein ≤ 70 g/L.
* Subject has screening serum albumin ≤ 38 g/L.

Exclusion Criteria:

* Subject is known to be allergic or intolerant to any ingredient found in the study product.
* Subject has pre-planned surgery other than hip fracture surgery during the study period.
* Subject has alcohol or substance abuse, severe dementia, brain metastases, eating disorders or any psychological condition that may interfere with dietary intake, severe nausea, vomiting, diarrhea, active gastritis, gastrointestinal bleeding or other gastrointestinal disturbances.
* Subject has active malignancy
* Subject has chronic, contagious, infectious disease, such as active tuberculosis, Hepatitis B or C, or HIV.
* Subject has diagnosis of IDDM.
* Subject has uncontrolled NIDDM determined by HbA1c > 8%.

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2009-11; Primary Completion 2010-08 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Blood chemistry | 28 days

SECONDARY OUTCOMES:
Product intake | 28 days
Functionality (pain, mobility, strength) | 28 days
Surgical site status | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Anne C Voss, PhD, Study Chair — Abbott Nutrition
Locations (11):
- Russia (11):
  - Regional Clinical Hospital #1, Krasnodar
  - City Clinical Hospital #15, Moscow
  - City Clinical Hospital #12, Moscow
  - City Clinical Hospital #31, Moscow
  - City Clinical Hospital n.a. Botkina, Moscow
  - State Novosibirsk Regional Hospital, Novosibirsk
  - Alexandrovskaya City Hospital, Saint Petersburg
  - Saint Petersburg State Medical Academy Mechnikova, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
  - Ufa Medical University, Hospital of Emergency Care, Ufa
  - Ural State Medical Academy, Yekaterinburg